CLINICAL TRIAL: NCT02365233
Title: A Phase IV, Open Label, Randomized Trial on the Effect of Metformin Plus Lantus Insulin, Pioglitazone, or DPP4 Inhibitor on Fatty Liver in Patients With Type II Diabetes
Brief Title: Fatty Liver Study in Patients With Type II Diabetes
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: IRB withheld the data due to inadequate supporting documentation
Sponsor: The University of Texas Medical Branch, Galveston (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 13-021
Record Dates: First submitted 2013-05-09; First posted 2015-02-18 (Estimated); Results first posted 2018-07-31 (Actual); Last update posted 2018-07-31 (Actual); Status verified 2018-04

CONDITIONS: Type II Diabetes; Nonalcoholic Fatty Liver
Keywords: Type II Diabetes; Nonalcoholic fatty liver
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Non-alcoholic Fatty Liver Disease | interventions — Dipeptidyl-Peptidase IV Inhibitors; saxagliptin; Pioglitazone; Insulin Glargine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Thiazolidinedione (Active Comparator): (Pioglitazone, 15 mg/day)
  Interventions: Drug: Pioglitazone
- Lantus Insulin (Active Comparator): 0.35 U per kg body weight once daily
  Interventions: Drug: Lantus insulin
- DPP4 inhibitor (Active Comparator): Sitagliptin, 100 mg/day or Saxagliptin, 5 mg/day
  Interventions: Drug: DPP4 inhibitor

INTERVENTIONS:
Drug: DPP4 inhibitor — Comparison between three common alternative therapeutic strategies to improve glycemic control in patients with type 2 diabetes who are not controlled with metformin alone.
  Other Names: sitagliptin100 mg daily; saxagliptin 5 mg daily
  Arms: DPP4 inhibitor
Drug: Pioglitazone — Comparison between three common alternative therapeutic strategies to improve glycemic control in patients with type 2 diabetes who are not controlled with metformin alone.
  Other Names: Pioglitazone 15 mg daily
  Arms: Thiazolidinedione
Drug: Lantus insulin — Comparison between three common alternative therapeutic strategies to improve glycemic control in patients with type 2 diabetes who are not controlled with metformin alone.
  Other Names: Lantus insulin (0.35U/kg of body weight once daily)
  Arms: Lantus Insulin

SUMMARY:
The primary objective of this trial is to measure changes in hepatic lipid content using three common alternative therapeutic strategies to improve glycemic control in patients with type 2 diabetes who are not controlled with metformin alone.

DETAILED DESCRIPTION:
In patients with type 2 diabetes whose glycemic control is not accomplished with Metformin alone, there are several options for additional hypoglycemic agent. As per recent National guidelines at least three "second line" agents can be added to metformin: thiazolidinediones, Lantus insulin, and DPP4 inhibitors. All three approaches have been proven to help accomplishing goals of therapy for glycemic control (HbA1c<7%) in clinical trials. Whether one approach is superior to the other in improving associated non-glycemic metabolic abnormalities and risk for future morbidity and mortality in patients with type 2 diabetes remains a matter of intense debate. Among these abnormalities, excessive triglyceride content in the liver (fatty liver or liver steatosis) is a major predictor of risk for non-alcoholic steato-hepatitis (NASH) and liver cirrhosis. Fatty liver is highly prevalent in patients with type 2 diabetes. There are no clinical studies done to determine if any of these three therapeutic options is superior at reducing the liver triglyceride content in patients with type 2 diabetes and fatty Liver. Therefore, in this study we propose to measure and compare the effects on liver triglyceride content when either pioglitazone, lantus insulin, or DPP4 inhibitors are added to metformin in patients with poorly controlled type 2 diabetes (HbA1c>7.6%) and fatty liver (presence of "bright" liver in abdominal ultrasound). The primary objective of this trial is to measure changes in hepatic lipid content using three common alternative therapeutic strategies to improve glycemic control in patients with type 2 diabetes who are not controlled with metformin alone.

ELIGIBILITY:
Inclusion Criteria:

1. Subject has provided informed consent in a manner approved by the Institutional Review Board (IRB) and is willing and able to comply with the trial procedures.
2. Adults at least 18 years of age at the time of consent.
3. Have type 2 diabetes mellitus.
4. Be on a stable medication with metformin (2000 mg/day) for at least 3 months prior to study enrollment.
5. Have blood A1c >7.6% and < 8.5% within 3 months prior to study enrollment.
6. Have fatty liver, which is diagnosed by ultrasonographic findings of "bright liver" within 1 year of study enrollment.
7. Stable medication for lipid lowering, blood pressure control, dietary supplements, including vitamins, for at least 3 months.
8. Women of Childbearing Potential must be willing and able to use acceptable forms of birth control while on the study.

Exclusion Criteria:

1. Currently taking medication that can affect glucose metabolism other than Metformin.
2. History of Kidney diseases that, in the opinion of the investigator , would place the subject at increased risk of participation or plasma levels of creatinine > 1.4 for women and > 1.5 for men.
3. History of Cirrhosis of liver, hepatitis, or other liver diseases that, in the opinion of the investigator, would place the subject at increased risk of participation.
4. Current alcohol consumption more than12 to 15 g of alcohol a day, or >12 oz of beer, 5 oz of wine, or 1.5 oz of distilled spirits.
5. History of heart failure.
6. Concurrent participation on another research study
7. Use of an investigational agent in the 30 days prior to signing informed consent.
8. History of prior non-compliance or the presence or history of psychiatric conditions (including drug or alcohol addiction) that would, in the opinion of the investigator, make it difficult for the subject to comply with the study procedures or follow the investigators instructions.
9. Females who are pregnant or lactating
10. Current Diagnosis or History of Bladder Cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2013-05-01 (Actual); Primary Completion 2016-12-31 (Actual); Study Completion 2016-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nicola Abate, MD, Principal Investigator — University of Texas Medical Branch-Galveston
Locations (1):
- University of Texas Medical Branch -Galveston, Galveston, Texas, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Before randomization to obtain the intervention, eligibility criteria were verified based on an A1c test, pregnancy test and liver ultrasound to confirm fatty liver.
  IRB withheld the data due to inadequate supporting documentation.
Period: Overall Study
Arm/Group | Thiazolidinedione | Lantus Insulin | DPP4 Inhibitor
Started | 1 | 2 | 2
Completed | 0 | 0 | 0
Not Completed | 1 | 2 | 2
Not completed — IRB withheld the data | 1 | 2 | 2

BASELINE CHARACTERISTICS:
Population: IRB withheld the data due to inadequate supporting documentation
Groups:
- Total: Total of all reporting groups
Arm/Group | Thiazolidinedione | Lantus Insulin | DPP4 Inhibitor | Total
Number analyzed (Participants) | 0 | 0 | 0 | 0
Age, Continuous [unit: years]
Sex: Female, Male

OUTCOME MEASURES:

1. Primary Outcome: Change in Hepatic Lipid Content From Baseline Visit to Six Month Follow up Visit
Description: Comparison of the hepatic lipid content measurement taken by MRI at baseline with the measurement taken by MRI at the 6 month follow up visit.
Time Frame: Hepatic lipid content measurement will be taken on Day #1 ( the day of randomization) and at the 6 month follow up visit.
Population: IRB withheld the data due to inadequate supporting documentation
Arm/Group | Thiazolidinedione | Lantus Insulin | DPP4 Inhibitor
Number analyzed (Participants) | 0 | 0 | 0
Statistical Analysis 1: Comparison: Thiazolidinedione vs Lantus Insulin vs DPP4 Inhibitor; Test type: Superiority; IRB withheld the data due to inadequate supporting documentation

ADVERSE EVENTS:
Description: IRB withheld the data due to inadequate supporting documentation
Arm/Group | Thiazolidinedione | Lantus Insulin | DPP4 Inhibitor
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
Inadequate documentation and lack of funding resulted in no usable data. IRB withheld the data.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No